CLINICAL TRIAL: NCT05562947
Title: A Phase III, Multicenter, Randomized, Visual Assessor-masked, Active-comparator Study of the Efficacy, Safety, and Pharmacokinetics of the Port Delivery System With Ranibizumab in Chinese Patients With Neovascular Age-related Macular Degeneration
Brief Title: A Study of the Efficacy, Safety, and Pharmacokinetics (PK) of the Port Delivery System With Ranibizumab (PDS) in Chinese Participants With Neovascular Age-related Macular Degeneration (nAMD)
Acronym: HUTONG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YR42983
Record Dates: First submitted 2022-09-15; First posted 2022-10-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Age-related Macular Degeneration; nAMD
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Implant Arm (Experimental): Participants will have the implant (pre-filled intraoperatively with ranibizumab 100 mg/mL) surgically inserted on Day 1. After Day 1, participants in the implant arm will attend monthly study visits, and receive implant refill-exchanges with ranibizumab 100 mg/mL at Week 24 and Week 48. At the Week 48 study visit, participants will move to the long -term extension phase of the study and continue receiving refill-exchanges Q24W until the end of study. Participants will attend monthly visits up to Week 96 and bi-monthly visits, thereafter.
  Interventions: Device: PDS With Ranibizumab (100 mg/mL)
- IVT Arm (Experimental): Participants will receive IVT ranibizumab 0.5 mg injections starting on Day 1. Participants will receive IVT ranibizumab 0.5 mg Q4W until Week 44. At the Week 48 study visit, participants will receive the PDS implant (pre-filled intraoperatively with ranibizumab 100 mg/mL), move to the long-term extension phase of the study and receive Q24W refill exchanges until the end of study. If participants are unable to attend the Week 48 visit due to extenuating circumstances, they should return no later than the next scheduled visit (Week 52), when they will receive the PDS implant. Participants will attend monthly visits up to Week 96 and bi-monthly visits, thereafter.
  Interventions: Drug: Ranibizumab (10 mg/mL)

INTERVENTIONS:
Device: PDS With Ranibizumab (100 mg/mL) — Participants randomized to the implant arm will have the implant (filled prior to implantation with approximately 20 microliters (μL) of the 100-mg/mL formulation of ranibizumab [approximately 2 mg dose of ranibizumab]) surgically inserted in the study eye at the Day 1 visit following their randomization visit, or at Week 48 visit for participants randomized to the IVT arm. After the initial fill of the implant with ranibizumab, participants will receive implant refill-exchanges at fixed 24-week intervals.
  Arms: Implant Arm
Drug: Ranibizumab (10 mg/mL) — Participants in the IVT arm will receive their first IVT injection of 50 μL of the 10 mg/mL ranibizumab (0.5 mg dose) at the Day 1 visit, which will occur at the conclusion of the randomization visit. Afterward, participants will receive IVT ranibizumab injections of 50 μL of the 10 mg/mL formulation Q4W at each scheduled study visit until Week 44.
  Arms: IVT Arm

SUMMARY:
This study will evaluate the efficacy, safety, and PK of ranibizumab 100 milligrams per milliliter (mg/mL) delivered every 24 weeks (Q24W) via the PDS implant compared with ranibizumab 0.5 milligrams (mg) delivered every 4 weeks (Q4W) as intravitreal (IVT) injection in chinese participants with nAMD.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of nAMD within 9 months prior to the screening visit
* Previous treatment with at least three anti-vascular endothelial growth factor (VEGF) IVT injections for nAMD per standard of care within 6 months prior to the screening visit
* Demonstrated response to prior anti-VEGF IVT treatment since diagnosis
* Availability of historical VA data prior to the first anti-VEGF treatment for nAMD up to the screening visit
* BCVA of 34 letters or better (20/200 or better approximate Snellen equivalent), using Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters
* All subtypes of nAMD lesions are permissible
* Sufficiently clear ocular media and adequate pupillary dilation to allow for analysis and grading by the central reading center of fundus photography (FP), fluorescein angiography (FA), indocyanine green angiography (ICGA), fundus autofluorescence (FAF), and optical coherence tomography (OCT) images

Exclusion Criteria:

A. Prior Ocular Treatment Study Eye

* History of vitrectomy surgery, submacular surgery, or other surgical intervention, all for AMD
* Prior treatment with Visudyne, external-beam radiation therapy, or transpupillary thermotherapy
* Previous treatment with corticosteroid IVT injection
* Previous intraocular device implantation (not including intraocular lens implants)
* Previous laser (any type) used for age-related macular degeneration (AMD) treatment
* Treatment with anti-VEGF agents other than ranibizumab within 1 month prior to the randomization visit
* Prior treatment with intravitreal treatments for geographic atrophy
* Concurrent conjunctival, Tenon's capsule, and/or scleral condition in the supero-temporal quadrant of the eye that may affect the implantation, subsequent tissue coverage, and refill-exchange procedure of the PDS implant

Either Eye

* Prior treatment with brolucizumab
* Prior gene therapy for nAMD or other ocular diseases
* Previous participation in any ocular disease studies of investigational drugs and/or devices, within 3 months or five elimination half-lives of the investigational therapy, whichever is longer, preceding the screening visit

B. Choroidal Neovascularization (CNV) Lesion Characteristics

Study Eye

* Subretinal hemorrhage that involves the center of the fovea, if the hemorrhage is greater than 0.5 disc area (1.27 millimeter square [mm^2]) in size at screening
* Subfoveal fibrosis or subfoveal atrophy

Either Eye • CNV due to other causes, such as ocular histoplasmosis, trauma, central serous chorio-retinopathy, or pathologic myopia

C. Concurrent Ocular Conditions Study Eye

* Retinal pigment epithelial tear
* Any concurrent intraocular condition
* Active intraocular inflammation (grade trace or above)
* History of vitreous hemorrhage
* History of rhegmatogenous retinal detachment
* History of rhegmatogenous retinal tears or peripheral retinal breaks within 3 months prior to the randomization visit
* History of pars plana vitrectomy surgery
* Aphakia or absence of the posterior capsule
* Spherical equivalent of the refractive error demonstrating more than 8 diopters of myopia
* Preoperative refractive error that exceeds 8 diopters of myopia, for participants who have undergone prior refractive or cataract surgery
* Intraocular surgery (including cataract surgery) within 3 months preceding the randomization visit
* Uncontrolled ocular hypertension or glaucoma
* History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery
* History of corneal transplant

Fellow (Non-Study) Eye

• Non-functioning fellow eye

Either Eye

* Any history of uveitis
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-07-27 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Best-corrected Visual Acuity (BCVA) Score Averaged Over Weeks 36 and 40, as Assessed Using the ETDRS Visual Acuity (VA) Chart at a Starting Distance of 4 Meters | Baseline up to Week 40

SECONDARY OUTCOMES:
Change From Baseline in BCVA Score Over Time | Baseline up to Week 144
Proportion of Participants With BCVA Score of 38 Letters (20/200 Approximate Snellen Equivalent) or Worse Averaged Over Weeks 36 and 40 | Baseline up to Week 40
Proportion of Participants With BCVA Score of 38 Letters (20/200 Approximate Snellen Equivalent) or Worse Averaged Over Weeks 44 and 48 | Baseline up to Week 48
Proportion of Participants With BCVA Score of 69 Letters (20/40 Approximate Snellen Equivalent) or Better Averaged over Weeks 36 and 40 | Baseline up to Week 40
Proportion of Participants With BCVA Score of 69 Letters (20/40 Approximate Snellen Equivalent) or Better Averaged Over Weeks 44 and 48 | Baseline up to Week 48
Proportion of Participants Who Gain ≥0 Letters in BCVA Score From Baseline Averaged Over Weeks 36 and 40 | Baseline up to Week 40
Proportion of Participants Who Gain ≥ 0 Letters in BCVA Score From Baseline Averaged Over Weeks 44 and 48 | Baseline up to Week 48
Proportion of Participants Who Lose < 10 or < 5 Letters in BCVA Score From Baseline Averaged Over Weeks 36 and 40 | Baseline up to Week 40
Proportion of Participants Who Lose < 10 or < 5 Letters in BCVA Score From Baseline Averaged Over Weeks 44 and 48 | Baseline up to Week 48
Change From Baseline in Center Point Thickness (CPT) at Week 36 | Baseline, Week 36
  CPT is retinal thickness in the center point of the fovea measured between the internal limiting membrane and the inner third of the retinal pigment epithelium layer. CPT will be measured using optical coherence tomography (OCT).
Change From Baseline in Central Subfield Thickness (CST) at Week 36 | Baseline, Week 36
  CST is defined as the average thickness of the central 1 millimeter (mm) circle of the ETDRS grid centered on the fovea. CST will be measured using OCT.
Change From Baseline in CPT at Week 44 | Baseline, Week 44
  CPT is retinal thickness in the center point of the fovea measured between the internal limiting membrane and the inner third of the retinal pigment epithelium layer. CPT will be measured using OCT.
Change From Baseline in CST at Week 44 | Baseline, Week 44
  CST is defined as the average thickness of the central 1 mm circle of the ETDRS grid centered on the fovea. CST will be measured using OCT.
Proportion of Participants in the Implant Arm Who do not Undergo Supplemental Treatment With IVT Ranibizumab 0.5 mg Before the First, Second, Third, Fourth, Fifth, and Sixth Fixed Refill-exchange Intervals | Baseline up to 144 weeks
Proportion of Participants in the Implant Arm Who do not Undergo a Supplemental Treatment that Requires Subsequent Additional Supplemental Treatments During the Study | Baseline up to 144 weeks
Percentage of Participants With Adverse Events (AEs) | Baseline up to 144 weeks
Percentage of Participants With Adverse Events of Special Interest (AESIs) | Baseline up to 144 weeks
Percentage of Participants With Ocular AESIs During the Post-operative Period and Follow-up Period | Post-operative period: up to 37 days after initial implantation Follow-up period: > 37 days after implantation surgery (up to 144 weeks)
Percentage of Participants Who Received PDS Affected With Adverse Device Effects (ADEs) | Baseline up to 144 weeks
Percentage of Participants Who Received PDS Affected With Anticipated Serious Adverse Device Effects (ASADEs) | Baseline up to 144 weeks
Number of Device Deficiencies | Baseline up to 144 weeks
Observed Serum Ranibizumab Concentrations at Specified Timepoints | Baseline, Weeks 4, 12, 24, 28, 36, 48
Area Under the Concentration Time Curve From 0-24 Weeks | Baseline, Weeks 4, 12, 24
Maximum Serum Concentration of Ranibizumab | Baseline, Weeks 4, 12, 24, 28, 36, 48
Minimum serum concentration of ranibizumab | Baseline, Weeks 4, 12, 24, 28, 36, 48
Number of Participants With Anti-drug Antibodies (ADAs) | Baseline, Weeks 4, 24, 48
Number of Participants With Treatment-emergent ADAs During the Study | Baseline, Weeks 4, 24, 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- China (16):
  - Peking Union Medical College Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - Qingdao Eye Hospital of Shandong First Medical University, Qingdao
  - Shanghai First People's Hospital, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - The First Affiliated Hospital of China Medical University, Shenyang
  - Shanxi Eye Hospital, Taiyuan
  - Tianjin Medical University Eye Hospital, Tianjin
  - Eye Hospital, Wenzhou Medical University, Wenzhou
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Xi'an People's Hospital (Xi'an Fourth Hospital), Xi'an

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing